CLINICAL TRIAL: NCT06894407
Title: Intra-tumoral Targeted Hyperthermic Therapy (THT) for Stage 3C/3D/4M1 Cutaneous Metastatic Melanoma in Patients with Targetable Cutaneous And/or Sub-cutaneous Tumors
Brief Title: Intratumoral Targeted Hyperthermia Therapy (THT) for Stage 3C/3D/4M1 Cutaneous Metastatic Melanoma
Acronym: THT-CMM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sona Nanotech Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP001
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cutaneous Metastatic Melanoma
Keywords: Hyperthermia; Gold Nanorods; Targeted Hyperthermia; Cutaneous Metastatic Melanoma Treatment; Near Infrared Light; Immunotherapy
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Targeted Hyperthermia Therapy (Experimental)
  Interventions: Device: Device: Targeted Hyperthermia Therapy

INTERVENTIONS:
Device: Device: Targeted Hyperthermia Therapy — Intra-tumoral gold nanorods (SivaRods) exposed to Near Infrared Light (860 +/- 10nm) mediated targeted hyperthermia therapy.
  Other Names: Gold Nanorods; Gold Nanoparticles

SUMMARY:
This phase I/II device clinical trial investigates the safety and efficacy of GNR-mediated THT in patients with stage 3C/3D/4M1 cutaneous metastatic melanoma unresponsive to systemic checkpoint immunotherapy or in patients who have contraindications to systemic immunotherapy.

The primary objective of the study is to evaluate the safety of THT treatment, with secondary objectives focused on tumor response to treatment.

Patients will receive intra-tumoral GNR injections, followed by NIR light therapy to induce mild hyperthermia, with intra-tumoral temperatures monitored to achieve a target range of 42°C to 48°C. The trial aims to establish a safe, effective dose of GNRs for THT therapy for cutaneous metastatic melanoma treatment and explore the potential for its localized tumor destruction.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older
* Participants with histologically or cytologically confirmed stage 3C/3D/4M1 advanced or cutaneous metastatic melanoma, with measurable disease by iRECIST including any number of cutaneous lesions
* Present a visible and accessible primary tumor or metastatic deposit (any site) that has not been surgically removed
* Present target tumors of 0.5 -2.5 cm in diameter
* Participants must have received and failed systemic and local intra-tumoral therapy at least one prior standard therapy, including immune checkpoint inhibitors (e.g., anti- PD1 or anti-CTLA-4), and failed local intra-tumoral IL-2 treatment. Failed response to treatment will be categorized according to iRECIST guidelines.
* Participants who have:

  * Immune partial response (iPR): At least a 30% decrease in the sum of diameters of target lesions compared to baseline, no progression of non-target lesions, No new lesions
  * Immune Stable Disease (iSD): Neither sufficient reduction to qualify for iPR nor sufficient increase to qualify for iCPD (immune confirmed progressive disease), no new lesions
  * Immune Unconfirmed Progressive Disease (iUPD); At least a 20% increase in the sum of diameters of target lesions, taking the smallest sum on study as the reference, appearance of new lesions, iUPD needs confirmation after at least 4 weeks; if confirmed, it becomes iCPD
  * Immune Confirmed Progressive Disease (iCPD): iUPD must be confirmed in a follow-up assessment (minimum of 4 weeks after initial iUPD), if progressive disease (increase in lesion size or additional new lesions) is still evident upon re-evaluation, iCPD is confirmed.
* Participants must agree to discontinue treatment with local intralesional immunotherapies during the study, with resumption after completion of the trial
* ECOG Performance Status:
* Life expectancy: ≥6 months
* Participants able and willing to provide written informed consent and comply with the trial protocol. 10. Either BRAF positive (BRAF+) or BRAF negative (BRAF-)

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the study.
* Women of childbearing potential must have a negative pregnancy test within 72 hours prior to enrollment and agree to use adequate contraception throughout the study
* Any infection requiring systemic therapy or other concurrent medical conditions (e.g., hepatitis B, hepatitis C, HIV) that would interfere with the study
* Myocardial infarction or stroke within the past 6 months, uncontrolled angina, or significant arrhythmia
* Participants receiving blood thinners as part of therapeutic anticoagulation therapy
* Any severe or uncontrolled comorbid condition that, in the investigator's opinion, would pose excessive risk to the participants (e.g., immunodeficiencies, severe hypertension, uncontrolled diabetes, liver failure)
* Participation in another clinical trial involving an investigational product/device within 30 days prior to screening
* Any condition that would impede compliance with study procedures
* Participants with a known allergy to gold of any kind
* Participants who are unable to tolerate cutaneous injections for any reason will not be eligible
* Participants with a known allergy to injectable local analgesics
* Participants with ocular melanoma or melanoma involving periorbital skin.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants that successfully complete THT (maintain intra-tumoral temperatures of 42-48C) | 1 year
  Total number of participants that successfully complete targeted hyperthermia therapy ie. maintain an intra-tumoral temperatures between 42-48C for 5 minutes
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 1 year
  The total number of participants experiencing adverse events, including serious adverse events, will be monitored and graded according to NCI CTCAE v5.0
Number of participants that have a tumor response as assessed by iRECIST 1.1 criteria | 1 year
  The total number of participants that have a tumor response to targeted hyperthermia therapy as assessed by iRECIST 1.1 criteria

SECONDARY OUTCOMES:
Number of participant's that have an increase in immune cell infiltrates in the tumor biopsy and blood samples post THT compared to pre-treatment patient samples | 1 year
  The total number of participants that have an increase in immune cell infiltrates in their tumor biopsy and blood samples following targeted hyperthermia therapy compared to patients biopsy and blood samples obtained before treatment

IPD SHARING:
Plan to Share IPD: Yes